CLINICAL TRIAL: NCT05556252
Title: The Effect of Hydrogen-rich Water Consumption on Premenstrual Symptoms and Quality of Life in Students With Premenstrual Syndrome: A Randomized Controlled Study
Brief Title: The Effect of Hydrogen-rich Water on Premenstrual Symptoms and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0720
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Hydrogenated water consumption
- Control Group (Placebo Comparator)
  Interventions: Other: Drinking water consumption

INTERVENTIONS:
Other: Hydrogenated water consumption — Participants will start consuming hydrogenated water on the 16th day of the menstrual cycle and will continue to apply it until the 2nd day of the next cycle. Within the scope of the study, they will be asked to drink of 300-400 ml hydrogenated water each morning before breakfast; 300-400 ml an hour before lunch; 300-400 ml two hours after lunch; 300-400 ml an hour before dinner; 300-400 ml half an hour before going to bed. Participants will be asked to consume a minimum of 1500 ml (1.5 L) and a maximum of 2000 ml (2.0 L) hydrogenated water in total. In this way, participants will be provided with hydrogenated water for three cycles.
  Arms: Intervention Group
Other: Drinking water consumption — Participants will start consuming drinking water on the 16th day of the menstrual cycle and will continue to apply it until the 2nd day of the next cycle. Within the scope of the study, they will be asked to drink of 300-400 ml drinking water each morning before breakfast; 300-400 ml an hour before lunch; 300-400 ml two hours after lunch; 300-400 ml an hour before dinner; 300-400 ml half an hour before going to bed. Participants will be asked to consume a minimum of 1500 ml (1.5 L) and a maximum of 2000 ml (2.0 L) drinking water in total. In this way, participants will be provided with drinking water for three cycles.
  Arms: Control Group

SUMMARY:
The aim of this study is to determine the effect of hydrogenated water on premenstrual symptoms and quality of life in students with premenstrual syndrome.

Research Hypotheses H1 1 Hydrogenated water consumption reduces premenstrual symptoms in students with premenstrual syndrome.

H1 2 Hydrogenated water consumption increases the quality of life in students with premenstrual syndrome.

The research will consist of intervention and control groups. Individuals consuming hydrogen-rich water will be included in the intervention group, whereas individuals consuming normal water will be in the control group. The block randomization method will be used to randomly assign participants who meet the research criteria to the groups. Participants will be provided with hydrogenated water for three cycles.

ELIGIBILITY:
Inclusion Criteria:

* The length of the menstrual cycle is within normal limits (21-35),
* Getting a score of 132 or more from the Premenstrual Syndrome Scale,
* Not receiving medical treatment for PMS,
* Not having any psychiatric diagnosis.

Exclusion Criteria:

* • Irregular menstruation in the last three cycles

  * Having received a psychiatric diagnosis,
  * Having any gynecological disease (abnormal uterine bleeding, myoma, ovarian cyst, etc.)
  * Using contraceptive medication.
  * Individuals' refusal to participate in the study,
  * Participants' non-compliance with the research plan,
  * Participants start receiving PMS treatment during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Change in premenstrual symptoms assessed by The Premenstrual Syndrome Scale | immediately before the intervention, immediately after the intervention, and 1 month after the intervention
  The Premenstrual Syndrome Scale (PMSS) consists of 44 questions. The PMSS is Likert type and its items are scored between 1 and 5 points. Lowest points of 44 and highest points of 220 can be obtained on the PMSS. The scale has a total of 9 subscales: depressive feeling, anxiety, fatigue, irritability, depressive thoughts, pain, changes in appetite, changes in sleeping habits and swelling. A higher score on the scale indicates that the severity of premenstrual syndrome is high.
Change in quality of life assessed by World Health Organization Quality of Life | immediately before the intervention, immediately after the intervention, and 1 month after the intervention
  The brief version of the World Health Organization Quality of Life (WHOQOL-BREF) is a sound, cross-culturally valid assessment of health-related quality of life in adults populations. Its assessment shows good to excellent internal consistency, test-retest reliability, discriminant validity, content validity, and construct validity in the healthy population and in different patient groups. Each question is scored from 1 to 5, with scores ranging from 0-100. A higher score means better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Nursing, Altindağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No